CLINICAL TRIAL: NCT07049354
Title: The Impact Of Media, Socioeconomic And Psychological Factors On The Adoption Of Aesthetic Technology And Cosmetic Surgery Among Women In Punjab, Pakistan
Brief Title: The Impact Of Media, Socioeconomic And Psychological Factors, Adoption Of Aesthetic Technology & CS
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/912
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Psychology, Social

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"This study titled "The Impact of Media, Socioeconomic and Psychological Factors on the Adoption of Aesthetic Technology and Cosmetic Surgery Among Women in Punjab, Pakistan" explores how various external and internal influences affect Pakistani women's decisions to undergo cosmetic procedures. With the rising trend of aesthetic treatments driven by modern beauty standards and social media exposure, the study investigates how psychological motivations, economic conditions, and media content shape these decisions. The increasing accessibility of non-invasive cosmetic options has made such procedures more common across different socio-economic groups.

DETAILED DESCRIPTION:
The research employs a cross-sectional survey and targets women aged 18-50 in urban and semi-urban areas of Lahore, Faisalabad, and Multan. A sample of 130 participants is selected using convenience sampling.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 50 years.
* Permanent residents of Punjab, Pakistan.
* Active users of social media platforms such as Instagram, TikTok, and Facebook.
* Regular consumers of cosmetic or beauty-related content on social media (e.g., following beauty influencers, engaging with posts about aesthetic procedures)

Exclusion Criteria:

* Participants will be excluded if they:
* Do not use social media.
* Fall outside the 18-50 age range.
* Have professional affiliations with the cosmetic industry, including cosmetic surgeons, beauty product marketers, or aesthetic practitioners, to minimize potential bias.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study employs a cross-sectional survey method to assess how media exposure, psychological motivations, and socio-economic factors influence the adoption of cosmetic surgery and aesthetic technologies among women in Punjab, Pakistan. A total of 130 women, aged 18 to 50, from Lahore, Faisalabad, and Multan were selected using convenience sampling. Data was collected through a structured and validated questionnaire covering demographics, media engagement, financial status, and self-perception.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
self administered questioner | 12 Months
  self administered quesioner with catogerical values to access the physocological stress

CONTACTS AND LOCATIONS:
Locations (1):
- Urban and semi-urban areas, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No